CLINICAL TRIAL: NCT06185725
Title: Comparison of Modified Perichondral Approach Thoracoabdominal Nerve Block and Transversus Abdominal Plane Block in Analgesia Management Following Caesarean Section Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Collaborators: Ahmet Kaciroglu (Unknown)
Responsible Party: Principal Investigator, Mursel Ekinci, Assoc prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 4
Record Dates: First submitted 2023-12-13; First posted 2023-12-29 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cesarean Section
Keywords: Cesarean Section Pain; Postoperative Analgesia; Transversus Abdominal Plane Block; Modified Perichondral Approach Thoracoabdominal Nerve Block

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Modified Perichondral Approach Thoracoabdominal Nerve block (M-TAPA block) group, and Transversus Abdominal Plane Block (TAP block) group
Who Masked: Participant, Outcomes Assessor
Masking Description: he patient and the outcomes assessor who performs postoperative pain evaluation will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA (Modified Perichondral Approach Thoracoabdominal Nerve block group) (Active Comparator): Patients will be performed to block at the end of the surgery. Patients will be administered paracetamol 1 gr (PERFALGAN® ) IV every 8 hours in the postoperative period.. If the patient's NRS score is ≥ 4 0,5 mg/kg IV meperidine (Aldolan ampul 100 mg/2 ml) will be administered.
  Interventions: Other: Modified Perichondral Approach Thoracoabdominal Nerve Block
- Group TAP (Transversus Abdominal Plane block group) (Active Comparator): Patients will be performed to block at the end of the surgery. Patients will be administered paracetamol 1 gr (PERFALGAN® ) IV every 8 hours in the postoperative period.. If the patient's NRS score is ≥ 4 0,5 mg/kg IV meperidine (Aldolan ampul 100 mg/2 ml) will be administered.
  Interventions: Other: Transversus Abdominal Plane Block

INTERVENTIONS:
Other: Modified Perichondral Approach Thoracoabdominal Nerve Block — M-TAPA block will be performed to Group M-TAPA at the end of the surgery, using US (Vivid Q) while the patient is in the supine position After providing aseptic conditions, the high frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The US probe will be placed in the sagittal plane where the midclavicular line intersects with the costal cartilage corresponding to the costochondral angle. Using the In Plane technique, the probe is gently pushed to visualize the lower part of the costochondral angle at the central level, advancing the block needle in the caudal-cranio direction, 5 ml of saline will be injected into the layer between the transverse abdominal muscle and the lower plane of the costal cartilage, and the block location will be confirmed. After the block location is confirmed, a total of 20 ml + 20 ml of 0.25% bupivacaine (total 40 ml for both sides) will be injected bilaterally
  Other Names: Postoperative analgesia management
  Arms: Group M-TAPA (Modified Perichondral Approach Thoracoabdominal Nerve block group)
Other: Transversus Abdominal Plane Block — TAP block will be performed to Group TAP at the end of the surgery, using US (Vivid Q) while the patient is in the supine position. After providing aseptic conditions, the high frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. USG will be placed transversely on the mid-axillary line between the iliac crest and subcostal planes. Using the In Plane technique, the block needle will be advanced into the fascial plane between the internal oblique and transversus abdominis muscles and the location will be confirmed by administering 5 ml of saline. The block needle will be advanced into the fascial plane between the internal oblique and transversus abdominis muscles and the location will be confirmed by administering 5 ml of saline.and than 20 ml of 0.25% bupivacaine (total 40 ml for both sides) will be injected bilaterally
  Other Names: Postoperative analgesia management
  Arms: Group TAP (Transversus Abdominal Plane block group)

SUMMARY:
Cesarean section (CS) is one of the most frequently performed surgical procedures in the World. Moderate to severe postoperative pain occurs in a significant proportion of women after cesarean surgery.

The analgesic effectiveness of TAP block has been demonstrated after cesarean section operations. m-TAPA block has been described as an alternative analgesic technique in abdominal surgeries.

The aim of this study is to compare these two analgesic methods in terms of effectiveness for postoperative analgesia management after cesarean section.

DETAILED DESCRIPTION:
Cesarean section (CS) is one of the most frequently performed surgical procedures in the World. In European countries, approximately 20% of deliveries are done by cesarean section. Moderate to severe postoperative pain occurs in a significant proportion of women after cesarean surgery. This delays recovery and returning to daily life. Postoperative pain disrupts the mother-child bond, makes breastfeeding difficult, and affects the psychological state of the mother.

Postoperative pain is an acute pain accompanied by the inflammatory process that occurs due to surgical trauma. Also inadequate postoperative analgesia may cause hyperalgesia and chronic pain. Perioperative pain should be managed with a multi-modal approach. Opioids and nonsteroid anti inflammatory drugs should be considered as components of a multimodal analgesic regimen. However, use of both systemic and neuraxial opioids may be associated with effects (respiratory depression, nausea, vomiting, sedation, pruritus, hyperalgesia). For this, interfacial blocks may be preffered to provide postoperative analgesia and reduced opioid consumption.

Regional analgesia techniques are performed as an important part of multimodal analgesia. US-guided Transversus abdominis plane (TAP) block is one of the regional analgesia techniques that can be performed preoperatively or postoperatively. TAP block has been shown to reduce postoperative pain after hysterectomy, inguinal hernia repair, cesarean section, and colorectal surgery.

Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block performed with ultrasound (US) is a novel technique that provides effective analgesia in the anterior and lateral thoracoabdominal areas, where local anesthetic is performed only to the lower side of the perichondral surface. M-TAPA block is a good alternative for analgesia of the upper dermatome levels and the abdominal lateral Wall, provides analgesia in the abdominal area at the T5-T11 level. In the literature, there are studies investigating the effectiveness of M-TAPA block for post-operative pain management in bariatric surgery.

The analgesic effectiveness of TAP block has been demonstrated after cesarean section operations. m-TAPA block has been described as an alternative analgesic technique in abdominal surgeries. The aim of this study is to compare these two analgesic methods in terms of effectiveness for postoperative analgesia management after cesarean section. The primary outcome is to compare global recovery scores, the secondary outcome is to compare postoperative pain scores (NRS), to evaluate postoperative rescue analgesic (opioid) use and side effects (allergic reaction, nausea, vomiting) associated with opioid use in this study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification II
* Elective cesarean section, and gestational age above 37 weeks will be included

Exclusion Criteria:

* Bleeding diathesis
* Anticoagulant treatment
* Local anesthetics and opioid allergy
* Infection at the site of block
* Patients who do not accept the procedure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Global recovery scoring system (patient satisfaction scale) | The quality of recovery will be evaluated out of a total of 150 points according to the QoR-15 test to be applied at the portoperative 24th hour.
  We will use the Turkish version of Quality of Recovery / QoR-15 questionairre
  PART A How have you been feeling in the last 24 hours? (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent])
  1. Able to breathe easily
  2. Been able to enjoy food
  3. Feeling rested
  4. Have had a good sleep
  5. Able to look after personal toilet and hygiene unaided
  6. Able to communicate with
  7. Getting support from hospital doctors and nurses
  8. Able to return to work or usual home activities
  9. Feeling comfortable and in control
  10. Having a feeling of general well-being
      PART B Have you had any of the following in the last 24 hours? (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor])
  11. Moderate pain
  12. Severe pain
  13. Nausea or vomiting
  14. Feeling worried or anxious
  15. Feeling sad or depressed

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | The NRS scores of the patients will be evaluated at the postoperative 0, 2, 4, 8, 16, and 24 hours.
  Postoperative 24 hours period. Patients' pain scores will be questioned at 0, 2, 4, 8, 16 and 24 hours.
The use of rescue analgesia | Meperidine consumption will be recorded at the first 24 hours period postoperatively. (total mg dose)
  The need for rescue analgesia will be recorded at the first 24 hours period postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- T.C. Sağlık Bakanlığı Bursa Şehir Hastanesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Visser GHA, Ayres-de-Campos D, Barnea ER, de Bernis L, Di Renzo GC, Vidarte MFE, Lloyd I, Nassar AH, Nicholson W, Shah PK, Stones W, Sun L, Theron GB, Walani S. FIGO position paper: how to stop the caesarean section epidemic. Lancet. 2018 Oct 13;392(10155):1286-1287. doi: 10.1016/S0140-6736(18)32113-5. No abstract available. PMID 30322563
- [Background] Roofthooft E, Joshi GP, Rawal N, Van de Velde M; PROSPECT Working Group* of the European Society of Regional Anaesthesia and Pain Therapy and supported by the Obstetric Anaesthetists' Association. PROSPECT guideline for elective caesarean section: updated systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 May;76(5):665-680. doi: 10.1111/anae.15339. Epub 2020 Dec 28. PMID 33370462
- [Background] Gamez BH, Habib AS. Predicting Severity of Acute Pain After Cesarean Delivery: A Narrative Review. Anesth Analg. 2018 May;126(5):1606-1614. doi: 10.1213/ANE.0000000000002658. PMID 29210789
- [Background] Tulgar S, Senturk O, Selvi O, Balaban O, Ahiskalioglu A, Thomas DT, Ozer Z. Perichondral approach for blockage of thoracoabdominal nerves: Anatomical basis and clinical experience in three cases. J Clin Anesth. 2019 May;54:8-10. doi: 10.1016/j.jclinane.2018.10.015. Epub 2018 Oct 31. No abstract available. PMID 30388604
- [Background] Ohgoshi Y, Ando A, Kawamata N, Kubo EN. Continuous modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) for major abdominal surgery. J Clin Anesth. 2020 Mar;60:45-46. doi: 10.1016/j.jclinane.2019.08.031. Epub 2019 Aug 20. No abstract available. PMID 31442859
- [Background] Sutton CD, Carvalho B. Optimal Pain Management After Cesarean Delivery. Anesthesiol Clin. 2017 Mar;35(1):107-124. doi: 10.1016/j.anclin.2016.09.010. Epub 2016 Dec 12. PMID 28131114